CLINICAL TRIAL: NCT02982746
Title: Can a Person-centred-care Intervention Improve Health-related Quality of Life in Patients With Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: University of Gothenburgh
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Health Related Quality of Life
Keywords: Head and neck cancer; Person Centred Care; Health related quality of life; EORTC QLQ-C30; EORTC QLQ-C35
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- gPCC-G (Gothenburg Person Centred Care) Group (Experimental): gPCC-G Patients randomized to the intervention group were contacted and scheduled to attend a meeting at the oncology clinic with the nurse specialist in oncology
  Interventions: Other: gPCC (Gothenburg Person Centred Care)
- Control group (No Intervention): Control Group Patients randomized to the control group received usual care and return visits were scheduled according to the treatment procedure described under the previous heading and based on the Regional care program for patients with HNC. CG patients were recruited at the same time and in the same way as those in the intervention group

INTERVENTIONS:
Other: gPCC (Gothenburg Person Centred Care)
  Arms: gPCC-G (Gothenburg Person Centred Care) Group

SUMMARY:
At all of the follow-ups, including the worst period (between four and ten weeks), the intervention group reported higher scores than the control group, suggesting in this RCT that adopting the person-centred-care concept was a promising way to improve function and wellbeing in patients with HNC.

DETAILED DESCRIPTION:
Background: The incidence of head and neck cancer (HNC) is increasing slightly. HNC and its treatment may affect general domains of health-related quality of life (HRQoL) and provoke a variety of adverse symptoms and side effects, both during and after treatment. The objective of this study was to compare a person-centred care intervention in terms of HRQoL, disease-specific symptoms or problems, with traditional care as a control group for patients with HNC. Methods: The intervention and control groups comprised 54 and 42 patients, respectively. Outcome measures used were: the EORTC QLQ-C30 and the EORTC QLQ-C35. Both groups answered the questionnaires at baseline and after 4, 10, 18 and 52 weeks from start of treatment. The questionnaires' scores were compared between groups by using independent samples test (Student's t-test) and non-parametric test (Mann-Whitney U Test) for continuous variables. For categorical data, Fisher's exact test was used. Longitudinal data were analysed using repeated measures in covariance pattern models. Results: At baseline, the intervention and control groups were comparable in terms of medical and sociodemographic variables, clinical characteristics, HRQoL and disease-specific symptoms or problems. At all the follow-up points, even during the worst period for the patients, the person-centred-care group consistently reported higher scores than the control group. The differences were numerically but not always statistically significant. When using repeated measures in covariance pattern models, statistically significant results were found for HNC-specific problems, swallowing (p= 0.014), social eating (p=0.048) and feeling ill (p=0.021).

ELIGIBILITY:
Inclusion Criteria:

* Eligible for this study were patients diagnosed with HNC, older than 18 years and able to read and write Swedish and, in addition, suitable for outpatient treatment with chemo- and/or radiotherapy, either as primary treatment or in a postoperative setting.

Exclusion Criteria:

* Patients were excluded if they had a previous or concomitant malignancy or were diagnosed and treated for depression as stated in their medical record.
* In order to minimize the risk of bias, none of the patients were to be included if they were taking part in other research studies

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Health related quality of life EORTC QLQ-30 EORTC QLQ-35 | Baseline
Health related quality of life EORTC QLQ-30 EORTC QLQ-35 | Four weeks
Health related quality of life EORTC QLQ-30 EORTC QLQ-35 | 10 weeks
Health related quality of life EORTC QLQ-30 EORTC QLQ-35 | 18 weeks
Health related quality of life EORTC QLQ-30 EORTC QLQ-35 | 52 weeks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gyllensten H, Koinberg I, Carlstrom E, Olsson LE, Hansson Olofsson E. Economic evaluation of a person-centred care intervention in head and neck oncology: results from a randomized controlled trial. Support Care Cancer. 2019 May;27(5):1825-1834. doi: 10.1007/s00520-018-4436-2. Epub 2018 Aug 31. PMID 30171334
- [Derived] Hansson E, Carlstrom E, Olsson LE, Nyman J, Koinberg I. Can a person-centred-care intervention improve health-related quality of life in patients with head and neck cancer? A randomized, controlled study. BMC Nurs. 2017 Feb 21;16:9. doi: 10.1186/s12912-017-0206-6. eCollection 2017. PMID 28239295